CLINICAL TRIAL: NCT05020964
Title: Screening Plasma HER2 Amplication by Digital PCR in Advanced Breast Cancer Patients Treated With Trastuzumab and Pyrotinib
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Screening plasma HER2 amplication by Digital PCR in Advanced Breast Cancer Patients Treated With Trastuzumab and Pyrotinib., Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC1888
Record Dates: First submitted 2021-08-19; First posted 2021-08-25 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2021-08

CONDITIONS: Advanced Breast Cancer
MeSH Terms: interventions — Trastuzumab; pyrotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Arm (Experimental): Trastuzumab and Pyrotinib
  Interventions: Drug: Trastuzumab and Pyrotinib

INTERVENTIONS:
Drug: Trastuzumab and Pyrotinib — Trastuzumab: 3-week dosing regimen, The initial load dose was 8 mg/kg. Pyrotinib: 400 mg orally once daily, take it continuously, every 21 days as a cycle.
  Use until intolerable toxicity or disease progression occurs.

SUMMARY:
The hypothesis of this study is to discover the efficacy and safety of trastuzumab combined with pyrotinib in treating advanced breast cancer with HER2 positive, which is detected by digital PCR. It is a single-arm, multicenter phase II clinical study.

The purpose of this study is:

1. To explore the Response rate (RR) and progression-free survival(PFS) and safety of patients with recurrent metastatic breast cancer who received trastuzumab combined with pyrotinib in positive plasma HER2 amplification detected by digital PCR.
2. To explore the potential using of digital PCR in recurrent and metastatic breast cancer.

DETAILED DESCRIPTION:
The purpose of this study is:

1. To explore the Response rate (RR) and progression-free survival(PFS) and safety of patients with recurrent metastatic breast cancer who received trastuzumab combined with pyrotinib in positive plasma HER2 amplification detected by digital PCR.
2. To explore the potential using of digital PCR in recurrent and metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with recurrent or distant metastatic breast cancer whose primary tissue was negative for HER2 amplification, and newly diagnosed patients with stage IV breast cancer who were negative for HER2 amplification; All enrolled patients had previously received ≥ second-line therapy; Note: ① negative expression of HER2 refers to the primary tissue tested by IHC/FISH (clinical report), and the cell immunohistochemical staining intensity is 0,1 + or 2+, but negative by fluorescence in situ hybridization (FISH).
2. Age range 18-75, female;
3. Good physical strength: ECOG score 0-1;
4. Expected survival of more than 3 months;
5. The patient had no major organ dysfunction;Include: Routine blood The ANC acuity 1.5 x 109 / L;PLT acuity 90 x 109 / L;Hb 90 g/L or higher; Blood biochemical 1.5 x ULN TBIL or less;ALT and AST 2 x ULN or less;ALT and AST≤5×ULN in patients with liver metastases;BUN and Cr≤1.5×ULN and creatinine clearance ≥50 mL/min (Cockcroft-Gault formula); Heart colour to exceed LVEF 50% or higher;Fridericia adjusted QT interval (QTcF) for 12-lead electrocardiogram in men < 450 ms and in women < 470 ms.
6. Evaluable tumor lesions according to RECIST 1.1 criteria;
7. Voluntarily join the group, agree and sign the written informed consent.

Exclusion Criteria:

1. Patients who have previously received anti-HER2 therapy, or who have received a study drug or preparation/treatment (i.e., participating in another trial) within 4 weeks prior to enrollment;
2. Patients who are allergic to study drugs or unable to take them orally;Patients who refuse the medication regimen;
3. Serious dysfunction of vital organs (heart, liver, kidney);Clinically significant heart disease, i.e., New York Heart Association (NYHA) grade ⅲ - ⅳ heart failure or more severe congestive heart failure or severe arrhythmias requiring pharmacological intervention;Uncontrollable angina pectoris, uncontrolled arrhythmia or uncontrolled hypertension, myocardial infarction within 6 months as confirmed by electrocardiogram (ECG);Previous history of organ transplantation, splenectomy;
4. Patients with other malignancies, except for cured non-melanoma skin cancers, cervical carcinoma in situ and other tumors that have been cured for at least 5 years;
5. Pregnant and lactating women (women of childbearing age are subject to pregnancy tests), fertile women with positive baseline pregnancy tests, or women of childbearing age who are unwilling to use effective contraception throughout the study period.;
6. In the active period of other acute infectious diseases or chronic infectious diseases;
7. A history of uncontrolled epilepsy, central nervous system disease or mental disorder;
8. Persons with disabilities of consciousness and other legal capacity or legal capacity limited;
9. A known history of human immunodeficiency virus;
10. Other conditions that the investigator considers inappropriate for the patient to participate in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-08-20 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate(ORR) | up to 1 year after the last patient enrolled
  The ORR will be defined as the proportion of patients in the Efficacy Evaluable patient Set who achieve complete response (CR) and partial response (PR)

SECONDARY OUTCOMES:
Progression free survival(PFS) | up to 1 year after the last patient enrolled
  PFS will be defined as the time from first dose of study drug until documentation of disease progression or death from any cause
Incidence and Severity of adverse events | approximately 1.5 years
  hematologic, hepatotoxicity, Incidence of hypertension, Incidence of proteinuria

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Peng, Study Chair — Cancer Institute and Hospital, Chinese Academy of Medical Sciences